CLINICAL TRIAL: NCT06896617
Title: Impact of the Presence of the Corpus Luteum on Pregnancies Obtained Through Frozen Embryo Transfer(FET): a Prospective Randomized Controlled Study
Brief Title: Impact of the Presence of the Corpus Luteum on Pregnancies Obtained Through Frozen Embryo Transfer(FET)
Acronym: LUTI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-513600-33-00; 2024-513600-33-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-05; First posted 2025-03-26 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-02

CONDITIONS: Infertilities; Embryo Transfer
MeSH Terms: interventions — Estradiol; Progesterone; Chorionic Gonadotropin; Thyrotropin Alfa

STUDY DESIGN:
Intervention Model Description: Evaluates the two procedures to become pregnant under study in order to find differences. Two arms and one control group of spontaneous pregnacies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PC-FET (endometrial preparation with absence of CL) (Active Comparator): Pregnancies with absence of corpus luteum
  Interventions: Drug: Estradiol + Progesterone
- NC-FET (natural cycle FET, endometrial preparation with presence of CL) (Active Comparator): Pregnancies with presence of corpus luteum
  Interventions: Drug: Ovitrelle ( Hcg 250 mcg)
- Control Arm (No Intervention): Spontaneous pregnancies with no intervention

INTERVENTIONS:
Drug: Estradiol + Progesterone — Pregnancies with absence of corpus luteum(PC-FET)
  Arms: PC-FET (endometrial preparation with absence of CL)
Drug: Ovitrelle ( Hcg 250 mcg) — NC-FET(natural cycle FET, endometrial preparation with presence of CL)
  Arms: NC-FET (natural cycle FET, endometrial preparation with presence of CL)

SUMMARY:
In pregnancies achieved through programmed frozen embryo transfer cycle (PC-FET) and modified natural frozen embryo transfer (mNC-FET), to determine whether there are differences in endothelial and placental function, maternal cardiovascular function, fetal growth and fetal cardiovascular and cerebral programming and to assess whether there is an association between these differences and the plasma concentrations of the main secretion products of the Corpus Luteum (CL) with vasoactive and angiogenic action.

ELIGIBILITY:
Inclusion Criteria:

* Female patients 18- 37 years old (both included) at the time of oocyte retrieval and less than 41 years of age at the time of embryo transfer.
* Regular menstrual cycles between 24 and 35 days.
* Availability of cryopreserved blastocysts from own gametes
* Indication for single embryo transfer.
* Patients who will be included in the LUTI study are candidates for either of the two procedures under study, and will have no contraindications for either procedure.

Exclusion Criteria:

* Recurrent pregnancy loss (3 or more).
* Recurrent implantation failure in previous IVF treatments (3 or more unsuccessful embryo transfers). .
* Diagnosis of polycystic ovarian syndrome, diabetes mellitus, chronic arterial hypertension, maternal heart disease and autoimmune diseases (Systemic Lupus Erythematosus (SLE) or Antiphospholipid syndrome (APS)).
* Active treatment with aspirin, heparin or other anticoagulant therapy, antihypertensives or other drugs used to treat circulation or coagulation disorders .
* Indication for PGT (Preimplantation Genetic Testing).
* Multiple pregnancy.

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 334 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-11-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Maternal: Relaxin-2 plasma concentrations. | Up to 10 month
Fetal: Mitral annular plane systolic excursion (MAPSE) assessed by echocardiography. | Up to 10 month

SECONDARY OUTCOMES:
Angiogenic/vasoactive function of corpus luteum and placenta | Up to 10 month
plasma concentrations of VCAM-1 and endoglin. | Up to 10 month
Maternal endothelial function | Up to 10 month
Maternal echocardiography: cardiac output (L/min) | Up to 10 month
Fetal programming | Up to 10 month
  Cardiac: sphericity index, longitudinal and transverse heart diameter (mm).
Fetal programming | Up to 10 month
  Cerebral cortex development: Depth of parietooccipital, cingulate and calcarine sulci (mm) corrected by DBP x 100
Fetal growth | At 12 week of gestation
  Fetal crown-rump length (CRL)(cm)
Fetal growth | At 20, 28, 32, and 36 week of gestation.
  Biometry (mm)
Neonatal data | At Delivery
  Apgar 5' test(parameter/puntuation)
Placental study | At Delivery
  Pregnancy: location of placenta (anterior, posterior, lateral or previa) and signs of placenta accreta spectrum disorders. Anatomopathologycal study of the placenta: weight (fresh, gr.) and histopathology
Preconceptional parameters | Visit 0 (Baseline)
  Both parents: age(years)
Maternal Cardivascular Function | Up to 10 month
  Plasma NT-proBNP concentration(pg/mL)
left ventricular remodeling parameters and total vascular resistance (dyn/sec/cm5). | Up to 10 month
Fetal programming | Up to 10 month
  Transverse and longitudinal diameters and sphericity index of atria and ventricles(mm).
Fetal programming | Up to 10 month
  Tricuspid annular plane systolic excursion (TAPSE)(mm).
Fetal programming | Up to 10 month
  Tricuspid annulus tissue Doppler [E', A' and S' wave (cms/s)].
Fetal programming | Up to 10 month
  Isovolumetric relaxation time (IRT)(mL/mmHg)
Fetal growth | At 12 week of gestation
  Nuchal translucency (NT)(mm)
Fetal growth | At 12 week of gestation
  ductus venosus pulsatility index (DV-PI)(pencentile)
Fetal growth | At 12 week of gestation
  Mean uterine artery pulsatility index (mUt-PI)(percentile)
Fetal growth | At 20, 28, 32, and 36 week of gestation.
  Biparietal diameter (BPD)(cm)
Fetal growth | At 20, 28, 32, and 36 week of gestation.
  Head circumference (HC)(cm)
Fetal growth | At 20, 28, 32, and 36 week of gestation.
  Abdominal circumference (AC)(cm)
Fetal growth | At 20, 28, 32, and 36 week of gestation.
  Femoral length (FL)(mm)
Fetal growth | At 20, 28, 32, and 36 week of gestation.
  Estimated fetal weight (g) and centile.
Fetal growth | At 20, 28, 32, and 36 week of gestation.
  Doppler study of umbilical artery (UA) middle cerebral artery (MCA) and mUt-PI (percentile)
Fetal growth | At 20, 28, 32, and 36 week of gestation.
  Study of Fetal Limb Volume (FLV) by 3D-echo (ml)
Neonatal data | At Delivery
  Umbilical artery pH(range)
Neonatal data | At Delivery
  Birth weight(kg)
Preconceptional parameters | Visit 0 (Baseline)
  Both parents: ethnicity(descriptive)
Preconceptional parameters | Visit 0 (Baseline)
  Both parents: socioeconomic status(descriptive)
Preconceptional parameters | Visit 0 (Baseline)
  Both parents: education level(descriptive),
Preconceptional parameters | Visit 0 (Baseline)
  Both parents:
  BMI(cm/kg)
Preconceptional parameters | Visit 0 (Baseline)
  Both parents: chronic diseases(descriptive)
Preconceptional parameters | Visit 0 (Baseline)
  Both parents: smoking(yes/no)
Preconceptional parameters | Visit 0 (Baseline)
  Both parents: alcohol consumption(yes/No)
Preconceptional parameters | Visit 0 (Baseline)
  Both parents: illicit substance abuse(Yes/No).
Maternal Cardivascular Function | Up to 10 month
  Systolic, diastolic and mean arterial blood pressure(mmHg)
Maternal Cardivascular Function | Up to 10 month
  Carotid artery intima-media thickness(mm)

CONTACTS AND LOCATIONS:
Locations (1):
- Laura Burunat, Barcelona, Spain, Spain